CLINICAL TRIAL: NCT06514508
Title: A Phase Ⅲ, Randomized, Double-Blinded Study Evaluating the Safety and Efficacy of Combination Treatment of Motixafortide and G-CSF as Compared to Placebo and G-CSF for the Mobilization of Hematopoietic Stem Cells for Autologous Transplantation in Subjects With Multiple Myeloma
Brief Title: Mobilization of Stem Cells With Motixafortide (BL-8040) in Combination With G-CSF in Multiple Myeloma Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLS-020-31
Record Dates: First submitted 2024-07-10; First posted 2024-07-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motixafortide+G-CSF (Experimental)
  Interventions: Drug: Motixafortide+G-CSF
- Placebo+G-CSF (Placebo Comparator)
  Interventions: Drug: Placebo+G-CSF

INTERVENTIONS:
Drug: Motixafortide+G-CSF — Patients will receive the first dose of motixafortide (1.25 mg/kg) by subcutaneous (SC) injection on the evening of Day 4 (10 to 14 hours) prior to initiation of the first apheresis. A second dose of motixafortide can be administered 10 to 14 hours before a third apheresis, if necessary for patients who did not reach the goal of collection. Injections of G-CSF per standard of care.
  Other Names: BL-8040+G-CSF
  Arms: Motixafortide+G-CSF
Drug: Placebo+G-CSF — Patients will receive the first dose of placebo by subcutaneous (SC) injection on the evening of Day 4 (10 to 14 hours) prior to initiation of the first apheresis. A second dose of placebo can be administered 10 to 14 hours before a third apheresis, if necessary for patients who did not reach the goal of collection. Injections of G-CSF per standard of care.
  Arms: Placebo+G-CSF

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multi-center phase Ⅲ bridging clinical study designed to evaluate the efficacy, safety, and pharmacokinetic and pharmacodynamic profiles of Motixafortide (BL-8040) + G-CSF vs placebo + G-CSF mobilized hematopoietic stem cells for autologous transplantation in Chinese patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* (Limit: 15,000 characters)

  1. Patients must have a signed study informed consent prior to entering the study.
  2. Patients must be between the ages of 18 and 78 years.
  3. Diagnosis of active multiple myeloma (aMM) as defined by IMWG criteria.
  4. At least one week (7 days) from last induction cycle of combination/multi-agent chemotherapy (e.g. KRD [carfilzomib, lenalidomide, dexamethasone] or VRD [bortezomib, lenalidomide, dexamethasone]) or from last single agent chemotherapy (e.g. lenalidomide, pomalidomide, bortezomib, dexamethasone, etc) prior to the first dose of G-CSF for mobilization.
  5. Eligible for Autologous Hematopoietic stem cell transplantation according to the Investigator's discretion.
  6. The subjects should be in first or second CR (including CR and SCR) or PR (including PR and VGPR).
  7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
  8. Adequate organ function at screening.
  9. Female subjects must be of non-childbearing potential or, if of childbearing potential, must have a negative serum pregnancy test at screening and negative serum pregnancy test within 72 hours prior to G-CSF first administration. Women of childbearing potential (WOCBP) and male subjects with WOCBP partners must agree to use highly effective contraception method during the study period and within 90 days after the last study treatment.

Exclusion Criteria:

1. Previous history of autologous or allogeneic-HCT.
2. Failed previous HSC collections or collection attempts.
3. Taken any of the listed below concomitant medications, growth factors or stimulating agents within the designated washout period:

   1. Dexamethasone: 7 days
   2. Thalidomide: 7 days
   3. Lenalidomide: 7 days
   4. Pamolidomide: 7 days
   5. Bortezomib: 7 days
   6. Carfilzomib: 7 days
   7. G-CSF: 14 days
   8. GM-CSF or Neulasta®: 21 days
   9. Erythropoietin or erythrocyte stimulating agents: 30 days
   10. Eltrombopag, romiplostim or platelet stimulating agents: 30 days
   11. Carmustine (BCNU): 42 days/6 weeks
   12. Daratumumab or any other anti-CD38: 28 days
   13. Ixazomib: 7 day.
4. Received >6 cycles lifetime exposure to thalidomide or lenalidomide.
5. Received >8 cycles of alkylating agent combinations.
6. Received > 6 cycles of melphalan.
7. Received prior treatment with radioimmunotherapy (e.g. radionuclides).
8. Received prior treatment with venetoclax.
9. Plans to receive maintenance treatment within 60 days post- transplantation (e.g.lenalidomide, bortezomib, pomalidomide, thalidomide, carfilzomib, etc.).
10. Has received a live vaccine within 30 days of the planned start of G-CSF administration. Seasonal flu vaccines that do not contain live virus are permitted.
11. Known active CNS metastases or carcinomatous meningitis.
12. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to motixafortide, G-CSF, or other agents used in the study.
13. Has an active or uncontrolled infection requiring systemic therapy.
14. Has a known additional malignancy that is progressing or requires active treatment.
15. Is currently participating and/or receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
16. O2 saturation < 92% (on room air).
17. Personal history or family history of Long QT Syndrome or Torsade de Pointes.
18. History of unexplained syncope, syncope from an uncorrected cardiac etiology, or family history of sudden cardiac death.
19. Myocardial infarction, CABG, coronary or cerebral artery stenting and/or angioplasty, stroke, cardiac surgery, or hospitalization for congestive heart failure within 3 months, Angina Pectoris Class >2 or NYHA Heart Failure Class >2.
20. ECG at screening showing QTcF > 470 msec and/or PR > 280 msec.
21. Mobitz II 2nd degree AV Block, 2:1 AV Block, High Grade AV Block, or Complete Heart Block, unless the patient has an implanted pacemaker or implantable cardiac defibrillator (ICD) with backup pacing capabilities.
22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Is pregnant or breast feeding or expecting to conceive or women of childbearing potential unless consent to use two contraceptive methods or highly effective contraception, within the projected duration of the trial, starting with the Screening Visit through 90 days after the last dose of study drug.
24. Known human immunodeficiency virus (HIV) or active Hepatitis B (e.g., Hepatitis B Surface Antigen [HBsAg] reactive and HBV DNA>500 IU/mL or >2500 copies/mL) or Hepatitis C (e.g., Hepatitis C Virus [HCV] RNA [qualitative] is positive).
25. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients mobilizing ≥6.0 × 10^6 CD34+ cells/kg with up to 2 apheresis sessions | Up to day 6

SECONDARY OUTCOMES:
Proportion of patients who collect ≥2.0 × 10^6 CD34+ cells/kg in 1 apheresis session | Up to Day 5
Proportion of patients who collect ≥6.0 × 10^6 CD34+ cells/kg in 1 apheresis session | Up to Day 5
Number of CD34+ cells/kg collected | Up to Day 8
Maximum plasma concentration (Cmax) | Up to Day 8
Time from transplantation to neutrophil engraftment | Up to post transplantation Day 29
Time from transplantation to platelets engraftment | Up to post transplantation Day 29
Graft durability at 100 days post-transplantation | Up to post transplantation Day 100
  Graft durability is defined as maintenance of at least 2 of the following 3 criteria:
  * Platelet count ≥50 × 10^9/L without transfusion for at least 2 weeks.
  * Hemoglobin level ≥10 g/dL with no erythropoietin support or transfusions for at least 1 month.
  * Absolute neutrophil count (ANC) ≥1.0 × 10^9/L for 1 week.
Change from Baseline in peripheral blood CD34+ cell concentration | Up to Day 8
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to Day 38

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Harbin The First Hospital, Harbin, Hei Longjiang